CLINICAL TRIAL: NCT06584396
Title: EMPOwER: Evaluating Mechanical Properties of Post-Mastectomy Skin Flaps to Estimate Reconstruction Risks
Brief Title: Evaluating Mechanical Properties of Post-Mastectomy Skin Flaps to Estimate Reconstruction Risks, the EMPOWER Study
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Artidis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-0320; NCI-2023-05588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2023-0320 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo tissue collection during standard of care surgery, have their medical records reviewed, and complete questionnaires throughout the study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the skin and surrounding soft tissue that is removed during an implant reconstruction after a mastectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize the nanomechanical properties of the skin and adjacent soft tissue removed at the time of postmastectomy implant reconstruction.

OUTLINE: This is an observational study.

Patients undergo tissue collection during standard of care surgery, have their medical records reviewed, and complete questionnaires throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* * Age 18 and older

  * Female sex
  * Patient with history of mastectomy with tissue expander placement
  * Tissue expander in place at time of study enrollment
  * Patient plans to undergo surgery to exchange tissue expander for permanent breast implant within the next 3 months of signing the informed consent
  * Ability to understand and provide written informed consent in accordance with institutional policies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with history of mastectomy with tissue expander placement recruited from MD Anderson.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Nanomechanical properties of the skin and adjacent soft tissue | At time of surgery
  The nanomechanical properties will be presented as a histogram that describes the characteristics of the sample. For each skin sample, summary statistics including mean (median), standard deviation, skewness, and range, mode, etc. will be used to describe the nanomechanical properties. Wilcoxon rank sum test or Fisher's exact test will be used to study the association between the summarized nanomechanical properties and clinical factors or outcomes. Pearson correlation coefficients will be used to assess the strength of association between any two continuous variables. Logistic regression will be conducted to examine the effect of nanomechanical properties on the risk of implant loss or any complication after adjusting other clinical factors.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Smith, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States